CLINICAL TRIAL: NCT00004652
Title: Phase II Pilot Controlled Study of Short Vs Longer Term Pimozide (Orap) Therapy in Tourette Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Rochester (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/11760; URMC-418
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Tourette Syndrome
Keywords: Tourette syndrome; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Tourette Syndrome; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Pimozide

INTERVENTIONS:
Drug: pimozide

SUMMARY:
OBJECTIVES: I. Determine whether the time period between randomization and endpoint is longer in the short term pimozide therapy or longer term therapy in patients with Tourette syndrome.

II. Determine whether tic severity, medication side effects, academic performance and psychosocial functioning are better in the short term pimozide therapy or longer term pimozide therapy.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a combined open label and double blind randomized study.

Patients receive pimozide (open label) orally until a stable level of tic control is achieved and remains unchanged for at least 1 month.

Then, patients are randomized to one of two possible double blind treatments. In the short term pimozide group, patients receive pimozide over 2 weeks. Then, pimozide is gradually replaced by an inactive placebo within the following 10 weeks.

Patients in the long term pimozide group receive pimozide. Patients continue treatment for 12 months or until a worsening of tics or behavioral symptoms are present for which an increased dosage is required.

Patients who do not experience an exacerbation of tics requiring an increase in dosage are followed for 1 year from the date of entry.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- DSM-III-R criteria for Tourette syndrome Chronic motor tic disorder with tics sufficiently severe to require neuroleptic therapy --Prior/Concurrent Therapy-- No clonidine for at least 2 weeks or any neuroleptic (e.g., haloperidol, pimozide) within 3 months prior to study Stable dosage of other medications (e.g., antiobsessional, stimulant) for at least 3 months prior to and during study required

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Start 1993-02

CONTACTS AND LOCATIONS:
Overall Officials: Roger Kurlan, Study Chair — University of Rochester

REFERENCES:
- [Background] Short-term versus longer term pimozide therapy in Tourette's syndrome: a preliminary study. Neurology. 1999 Mar 10;52(4):874-7. doi: 10.1212/wnl.52.4.874. PMID 10078748